CLINICAL TRIAL: NCT01918761
Title: Dacomitinib + Pemetrexed for Patients With Advanced Non-squamous Non-small Cell Lung Cancer (NSCLC): a Phase I Trial to Identify a Dose of Dacomitinib in Combination With Pemetrexed That is Safe and Tolerated as Determined by the Incidence of Dose Limiting Toxicities (DLTs)
Brief Title: Dacomitinib + Pemetrexed for Patients With Advanced Non-squamous Non-small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Central European Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CECOG/ NSCLC.1.1.001
Record Dates: First submitted 2013-05-27; First posted 2013-08-08 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2018-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; Stage IV; Pemetrexed; Dacomitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dacomitinib, Pemetrexed (Experimental): Pemetrexed 500mg/m2 (i.v) q21d Dacomitinib 45mg/ orally (continuous)
  Interventions: Drug: Dacomitinib, Pemetrexed

INTERVENTIONS:
Drug: Dacomitinib, Pemetrexed — Pemetrexed 500mg/m2 i.v (q21d) Dacomitinib 45mg orally (continuous)
  Other Names: Alimta

SUMMARY:
To identify a dose of dacomitinib in combination with pemetrexed that is safe and tolerated as determined by the incidence of DLTs (dose limiting toxicities).

DETAILED DESCRIPTION:
This open label phase Ib trial aims to determine the safety, tolerability, the pharmacokinetic profile, and to identify a dose of dacomitinib in combination with pemetrexed.

Three sites in Austria will participate in this study. Six to nine patients will initially be enrolled to receive the target dose of 45 mg qd dacomitinib (starting from day 2 of first cycle) in combination with pemetrexed (500 mg/m² 10 min infusion, once every 3 weeks). One cycle is defined as 21 days.

The first 3 subjects will be enrolled at a rate of ≤ 1 subject per week. If the target dose regimen is safe based on the incidence of DLT another 3 subjects will be enrolled.

If the dose of 45 mg qd is not safe alternate lower doses will be explored (dose level -1, dose level -2) to identify the maximal tolerated dose (MTD) of dacomitinib in combination of pemetrexed. Six to nine patients per dose level will be enrolled.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* Histologically or cytologically confirmed stage IV non-squamous NSCLC
* Patients who are candidates to receive pemetrexed monotherapy
* If pemetrexed has been administered as first line therapy there must be a treatment free interval of at least one cycle (21 days)
* Measurable disease by RECIST criteria version 1.1.
* ≥18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Adequate left ventricular ejection fraction (LVEF) ≥ 50% by either echocardiogram or multigated acquisition scan (MUGA)
* Adequate organ function, including:

  1. Adequate bone marrow reserve: absolute neutrophil count (ANC) should be ≥ 1500 cells/mm3, platelets should be ≥ 100.000 cells/mm3
  2. Creatinine clearance ≥ 45 mL/min
  3. Total bilirubin ≤ 1.5 x upper normal limit (ULN)
  4. Aspartate Aminotransferase (AST) (SGOT) ≤ 3 x ULN (≤ 5.0 x ULN if hepatic metastases)
  5. Alanine Aminotransferase (ALT) (SGPT) ≤ 3 x ULN (≤ 5.0 x ULN if hepatic metastases)
* Female patients or their partners must be postmenopausal (defined as 12 months of amenorrhea following last menses), surgically sterile or must agree to use effective contraception while receiving trial treatment and for at least 3 months thereafter (the definition of effective contraception will be based on the judgment of the investigator). Male patients or their partners must be surgically sterile or must agree to use a barrier method of contraception while receiving trial treatment and for at least 3 months thereafter. (In all cases the definition of effective contraception will be based on the judgment of the investigator).
* Able to comply with required protocol procedures and able to receive oral medications

Exclusion criteria:

* Any evidence of mixed histology that includes elements of small cell or carcinoid lung cancer
* Predominantly squamous cell histology
* Patients with symptomatic brain metastases
* Chemotherapy, radiotherapy, biological or investigational agents within two weeks of baseline disease assessments
* Patients with uncontrolled or significant cardiovascular disease, including:

  1. Myocardial infarction within 12 months
  2. Uncontrolled angina within 6 months
  3. Congestive heart failure within 6 months
  4. Diagnosed or suspected congenital long QT syndrome
  5. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
  6. Prolonged QTc interval on pre-entry electrocardiogram. QTc must be less than CTC Grade 2 (≤480 msec) using appropriate correction formula with manual read by investigator if required. The echocardiogram (ECG) may be repeated for evaluation of eligibility after management of correctable causes for observed QTc prolongation
  7. Any history of second or third degree heart block (may be eligible if currently have a pacemaker)
  8. Heart rate <50/minute on baseline electrocardiogram
  9. Uncontrolled hypertension
* Prior malignancy: Patients will not be eligible if they have evidence of other malignancy (other than non-melanoma skin cancer or in situ cervical cancer, or localized and presumed cured prostate cancer with prostate specific antigen (PSA) < ULN) within the last 3 years.
* Pregnant or lactating females. Serum pregnancy test to be assessed within 7 days prior to study treatment start. Known hypersensitivity to pemetrexed and/or dacomitinib
* Patients with exposure to other investigational drug therapy
* Previous therapy with an oral tyrosine kinase inhibitor (TKI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-07-30; Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph C Zielinski, Univ. Prof., Principal Investigator — Univ Clinic for Internal Medicine I, Dep of Oncology, Medical University of Vienna
Locations (2):
- Austria (2):
  - Medizinische Universität Graz Klinische Abteilung für Onkologie, Graz
  - Universitätsklinik für Innere Medizin I, Innsbruck

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dacomitinib, Pemetrexed
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Dacomitinib, Pemetrexed
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/ Caucasian | 5
Region of Enrollment [Number; unit: participants]
  Austria | 5
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — 0 - Asymptomatic, 1 - Symptomatic but completely ambulatory, 2 - Symptomatic, <50% in bed during the day, 3 - Symptomatic, >50% in bed, but not bedbound, 4 - Bedbound, 5 - Death
  Participants
    0 | 4
    1 | 1
KRAS status [Count of Participants; unit: Participants]
  Negative | 1
  Not determined | 4
Epidermal growth factor receptor (EGFR) mutation status [Count of Participants; unit: Participants]
  Negative | 1
  Not determined | 4
Weight [Mean (Standard Deviation); unit: kg] | 73.8 (9.68)
Heart rate [Mean (Standard Deviation); unit: bpm] | 70.6 (8.62)
Height [Mean (Standard Deviation); unit: cm] | 176.4 (14.26)
Temperature [Mean (Full Range); unit: °C] | 36.4 [36.0 to 36.8]
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m²] | 1.9 (0.20)
Stage at primary diagnosis: Primary tumor (T) [Count of Participants; unit: Participants] — Tis - Carcinoma in situ, Tx - Primary Tumor cannot be assessed, T1b - Tumor > 10 mm but ≤ 20 mm in greatest dimension, T2a - Tumor > 30 mm but ≤ 40 mm in greatest dimension, T3 - Tumor > 50 mm but ≤ 70 mm in greatest dimension or tumor of any size with direct extension to chest wall, pericadium, phrenic nerve or satellite nodules in the same lobe, T4 - Tumor > 70 mm or any tumor with Invasion of mediastinum, diaphragm, heart, great vessels, recurrent laryngeal nerve, carina, trachea, oesophagus, spine or separate tumor in different lobe of ipsilateral lung
  Participants
    T0 | 1
    T1b | 1
    T2a | 2
    T4 | 1
Stage at primary diagnosis: Regional lymph nodes (N) [Count of Participants; unit: Participants] — Nx - Regional lymph nodes cannot be assessed, N0 - No regional lymph node metastases, N1 - Metastasis to ipsilateral peribronchial and/or hilar lymph nodes, N2 - Metastasis to ipsilateral mediastinal and/or subcarinal lymph nodes, N3 - Metastasis to scalene or supraclavicular lymph nodes, metastasis to contralateral hilar or mediastinal lymph nodes
  Participants
    N0 | 2
    N2 | 2
    N3 | 1
Stage at primary diagnosis: Distant metastasis (M) [Count of Participants; unit: Participants] — M0 - No clinical or radiographic evidence of distant metastases, M1 - Distant metastases detected, Mx - Metastases cannot be assessed.
  Participants
    M0 | 1
    M1 | 4
Prior chemotherapy [Count of Participants; unit: Participants]
  Yes | 5
  No | 0
Prior surgery [Count of Participants; unit: Participants]
  Yes | 5
  No | 0
Prior radiotherapy [Count of Participants; unit: Participants]
  Yes | 0
  No | 5
Prior antibody therapy [Count of Participants; unit: Participants]
  Yes | 0
  No | 5
Electrocardiogram (ECG) results [Count of Participants; unit: Participants]
  Abnormal | 1
  Normal | 4
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: percent] | 65.2 (12.28)

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLTs)
Description: The primary objective of this study is to determine the maximal tolerated dose (MTD) of the combination pemetrexed + dacomitinib by the incidence of dose limiting toxicities (DLTs).
Time Frame: From start of treatment to end of treatment or death, whichever occurs first. The study was suspended after 36 months.
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dacomitinib, Pemetrexed
Number analyzed (Participants) | 5
percentage of participants | 40 [5.3 to 85.3]

2. Secondary Outcome: Overall Response Rate
Description: Overall Response Rate (ORR) is defined as the proportion of patients with complete Response (CR) or partial Response (PR).
Time Frame: Until progression of disease (PD) or 24 month after end of treatment for participants with no PD. The study was suspended after 36 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dacomitinib, Pemetrexed
Number analyzed (Participants) | 5
percentage of participants | 0 [0 to 52.2]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) defined as time from start of Dacomitinib to date of death from any cause. Patients without recorded death were censored at the date the patient was last known to be alive. Patients were followed up for survival for 24 month after end of Treatment.
Time Frame: until date of death. The study was suspended after 36 months.
Population: All enrolled participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacomitinib, Pemetrexed
Number analyzed (Participants) | 5
months | 9.6 [2.7 to NA] — The upper confidence interval was not reached due to an insufficient number of events.

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) defined as time from start of Dacomitinib to date of progression or date of death from any cause, whichever occurred first. Patients without recorded progression or death were censored at the last date they were known to have not progressed. Patients were followed up for progression-free survival for 24 month after end of Treatment.
Time Frame: Up to progression or death due to any cause. The study was suspended after 36 months
Population: All enrolled participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacomitinib, Pemetrexed
Number analyzed (Participants) | 5
months | 4.7 [1.4 to NA] — The upper confidence interval was not reached due to an insufficient number of events.

ADVERSE EVENTS:
Time Frame: From first dose of the study drugs until the 28-day post-treatment follow up visit, up to approximately 36 months.
Arm/Group | Dacomitinib, Pemetrexed
All-Cause Mortality (participants affected / at risk) | 3/5
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dacomitinib, Pemetrexed (N=5)
Dyspnoea (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
General physical condition abnormal (Investigations) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dacomitinib, Pemetrexed (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 (6)
Neutropenia (Blood and lymphatic system disorders) | 1 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3)
Dyspnoea (Cardiac disorders) | 1 (1)
Eye infection (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Burning mouth syndrome (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (11)
Nausea (Gastrointestinal disorders) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 4 (5)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Polyneuropathy (Nervous system disorders) | 1 (1)
Symmetrical drug-related intertriginous and flexural exanthema (Immune system disorders) | 2 (6)
General physical condition abnormal (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (3)
White blood cell count decreased (Investigations) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2)
Weight loss poor (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (3)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 (1)
Paronychia (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Scrotal ulcer (Skin and subcutaneous tissue disorders) | 1 (3)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes